CLINICAL TRIAL: NCT04468009
Title: Treatment of Critically Ill Patients With Covid-19 With Convalescent Plasma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital de Infecciosas Francisco Javier Muniz (Other Government)
Responsible Party: Principal Investigator, Carlos Alberto Gonzalez, Blood Bank Director in Hospital de Infecciosas Francisco Javier Muniz, Hospital de Infecciosas Francisco Javier Muniz
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1725
Record Dates: First submitted 2020-07-09; First posted 2020-07-13 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: SARS-Associated Coronavirus; Covid19; SARS-CoV Infection
Keywords: Convalescent plasma; Covid-19 treatment; Transfusion medicine
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care (No Intervention): Standard of care for Covid-19
- PCC-19 (Experimental): Treatment with convalescent plasma
  Interventions: Biological: Convalescent plasma

INTERVENTIONS:
Biological: Convalescent plasma — Convalescent plasma from patients recovering from Covid-19 and which had anti-SARS-Cov-2 antibodies
  Arms: PCC-19

SUMMARY:
This study aims to collect convalescent plasma and use it as experimental treatment in critically ill Covid-19 patients in order to reduce mortality and length of stay in intensive care unit.

DETAILED DESCRIPTION:
This study aims to use convalescent plasma as experimental treatment in critically ill Covid-19 patients in order to reduce mortality and length of stay in intensive care unit. Donors must have anti-SARS CoV2 antibodies. Recipients must be critically ill Covid-19 patients on mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years or more.
* Patient with Covid-19 confirmed with nuclear acid testing
* Critically ill patients with Covid-19 on mechanical ventilation. Potencially critically ill patients (with acute respiratory distress syndrome, septic shock and/or multiple organ failure) with Covid-19.
* Diagnosed with acute respiratory distress syndrome.
* Informed consent.

Exclusion Criteria:

* No consent.
* Symptoms for a period longer than 20 days.
* Not detectable by acid nuclear testing within 48 hours prior to elegibility.
* Descompensated congestive heart failure, in which receiving 500ml of intrasvascular volume signifies a life risk.
* History of severe adverse events or anaphylaxis to plasma components

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2021-01-19 (Actual); Study Completion 2021-06-19 (Actual)

PRIMARY OUTCOMES:
Mortality at ICU at 30 days | Mortality at 30 days
  Mortality at 30 days of Intensive Care Unit (ICU) admission
Mortality at ICU at 90 days | Mortality at 90 days
  Mortality at 90 days of ICU admission

SECONDARY OUTCOMES:
SOFA score of study days 1, 3, 5, 7, 14 and 28 | Study days 1, 3, 5, 7, 14 and 28
  Sequential Organ Failure Assessment (SOFA) of study days 1, 3, 5, 7, 14 and 28
Need for supportive therapy after enrollment | Duration of supportive therapy through study completion, an average of 3 months
  Duration (number of days) of supportive therapy (oxygen and ventilation, dialysis, vasopressors) after enrollment
Lenght of stay in ICU | Duration of stay in ICU through study completion, an average of 3 months
  Duration (number of days) of stay in ICU between ICU admission and ICU final discharge
Lenght of mechanical ventilation | Duration of mechanical ventilation through study completion, an average of 3 months
  Duration (number of days) of mechanical ventilation between beginning and final liberation from mechanical ventilation
Lenght of hospitalization | Duration of hospitalization through study completion, an average of 3 months
  Duration (number of days) of hospitalization between hospital admission and final hospital discharge

OTHER OUTCOMES:
Lenght of hospitalization after ICU discharge | Duration (number of days) of hospitalization through study completion, an average of 3 months
  Duration (number of days) of hospitalization after ICU discharge
Days without ventilation after enrollment | Days without ventilation through study completion, an average of 3 months
  Number of days without ventilation after enrollment
Days without vasopressors after enrollment | Days without vasopressors through study completion, an average of 3 months
  Number of days without vasopressors after enrollment
Changes in Chest X-ray | Changes in Chest X-ray through study completion, an average of 3 months
  Changes in Chest X-ray (unilateral, bilateral, unique, multiple, pleural effusion) after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Gonzalez, MD, Principal Investigator — Hospital de Infecciosas Francisco Javier Muniz
Locations (1):
- Hospital Francisco Javier Muñiz, Ciudad Autonoma de Buenos Aire, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Enria DA, Briggiler AM, Fernandez NJ, Levis SC, Maiztegui JI. Importance of dose of neutralising antibodies in treatment of Argentine haemorrhagic fever with immune plasma. Lancet. 1984 Aug 4;2(8397):255-6. doi: 10.1016/s0140-6736(84)90299-x. PMID 6146809
- [Background] Rojas M, Rodriguez Y, Monsalve DM, Acosta-Ampudia Y, Camacho B, Gallo JE, Rojas-Villarraga A, Ramirez-Santana C, Diaz-Coronado JC, Manrique R, Mantilla RD, Shoenfeld Y, Anaya JM. Convalescent plasma in Covid-19: Possible mechanisms of action. Autoimmun Rev. 2020 Jul;19(7):102554. doi: 10.1016/j.autrev.2020.102554. Epub 2020 May 5. PMID 32380316
- [Background] Duan K, Liu B, Li C, Zhang H, Yu T, Qu J, Zhou M, Chen L, Meng S, Hu Y, Peng C, Yuan M, Huang J, Wang Z, Yu J, Gao X, Wang D, Yu X, Li L, Zhang J, Wu X, Li B, Xu Y, Chen W, Peng Y, Hu Y, Lin L, Liu X, Huang S, Zhou Z, Zhang L, Wang Y, Zhang Z, Deng K, Xia Z, Gong Q, Zhang W, Zheng X, Liu Y, Yang H, Zhou D, Yu D, Hou J, Shi Z, Chen S, Chen Z, Zhang X, Yang X. Effectiveness of convalescent plasma therapy in severe COVID-19 patients. Proc Natl Acad Sci U S A. 2020 Apr 28;117(17):9490-9496. doi: 10.1073/pnas.2004168117. Epub 2020 Apr 6. PMID 32253318
- [Background] Shen C, Wang Z, Zhao F, Yang Y, Li J, Yuan J, Wang F, Li D, Yang M, Xing L, Wei J, Xiao H, Yang Y, Qu J, Qing L, Chen L, Xu Z, Peng L, Li Y, Zheng H, Chen F, Huang K, Jiang Y, Liu D, Zhang Z, Liu Y, Liu L. Treatment of 5 Critically Ill Patients With COVID-19 With Convalescent Plasma. JAMA. 2020 Apr 28;323(16):1582-1589. doi: 10.1001/jama.2020.4783. PMID 32219428
- [Background] Zhang B, Liu S, Tan T, Huang W, Dong Y, Chen L, Chen Q, Zhang L, Zhong Q, Zhang X, Zou Y, Zhang S. Treatment With Convalescent Plasma for Critically Ill Patients With Severe Acute Respiratory Syndrome Coronavirus 2 Infection. Chest. 2020 Jul;158(1):e9-e13. doi: 10.1016/j.chest.2020.03.039. Epub 2020 Mar 31. PMID 32243945
- [Background] Ahn JY, Sohn Y, Lee SH, Cho Y, Hyun JH, Baek YJ, Jeong SJ, Kim JH, Ku NS, Yeom JS, Roh J, Ahn MY, Chin BS, Kim YS, Lee H, Yong D, Kim HO, Kim S, Choi JY. Use of Convalescent Plasma Therapy in Two COVID-19 Patients with Acute Respiratory Distress Syndrome in Korea. J Korean Med Sci. 2020 Apr 13;35(14):e149. doi: 10.3346/jkms.2020.35.e149. PMID 32281317
- [Background] Ye M, Fu D, Ren Y, Wang F, Wang D, Zhang F, Xia X, Lv T. Treatment with convalescent plasma for COVID-19 patients in Wuhan, China. J Med Virol. 2020 Oct;92(10):1890-1901. doi: 10.1002/jmv.25882. Epub 2020 Jun 29. PMID 32293713
- [Background] Rajendran K, Krishnasamy N, Rangarajan J, Rathinam J, Natarajan M, Ramachandran A. Convalescent plasma transfusion for the treatment of COVID-19: Systematic review. J Med Virol. 2020 Sep;92(9):1475-1483. doi: 10.1002/jmv.25961. Epub 2020 May 12. PMID 32356910
- [Background] Joyner M, Wright RS, Fairweather D, Senefeld J, Bruno K, Klassen S, Carter R, Klompas A, Wiggins C, Shepherd JR, Rea R, Whelan E, Clayburn A, Spiegel M, Johnson P, Lesser E, Baker S, Larson K, Ripoll Sanz J, Andersen K, Hodge D, Kunze K, Buras M, Vogt M, Herasevich V, Dennis J, Regimbal R, Bauer P, Blair J, van Buskirk C, Winters J, Stubbs J, Paneth N, Casadevall A. Early Safety Indicators of COVID-19 Convalescent Plasma in 5,000 Patients. medRxiv [Preprint]. 2020 May 14:2020.05.12.20099879. doi: 10.1101/2020.05.12.20099879. PMID 32511566
- [Background] Valk SJ, Piechotta V, Chai KL, Doree C, Monsef I, Wood EM, Lamikanra A, Kimber C, McQuilten Z, So-Osman C, Estcourt LJ, Skoetz N. Convalescent plasma or hyperimmune immunoglobulin for people with COVID-19: a rapid review. Cochrane Database Syst Rev. 2020 May 14;5(5):CD013600. doi: 10.1002/14651858.CD013600. PMID 32406927
- [Background] Mair-Jenkins J, Saavedra-Campos M, Baillie JK, Cleary P, Khaw FM, Lim WS, Makki S, Rooney KD, Nguyen-Van-Tam JS, Beck CR; Convalescent Plasma Study Group. The effectiveness of convalescent plasma and hyperimmune immunoglobulin for the treatment of severe acute respiratory infections of viral etiology: a systematic review and exploratory meta-analysis. J Infect Dis. 2015 Jan 1;211(1):80-90. doi: 10.1093/infdis/jiu396. Epub 2014 Jul 16. PMID 25030060
- [Background] Guo L, Ren L, Yang S, Xiao M, Chang D, Yang F, Dela Cruz CS, Wang Y, Wu C, Xiao Y, Zhang L, Han L, Dang S, Xu Y, Yang QW, Xu SY, Zhu HD, Xu YC, Jin Q, Sharma L, Wang L, Wang J. Profiling Early Humoral Response to Diagnose Novel Coronavirus Disease (COVID-19). Clin Infect Dis. 2020 Jul 28;71(15):778-785. doi: 10.1093/cid/ciaa310. PMID 32198501
- [Background] To KK, Tsang OT, Leung WS, Tam AR, Wu TC, Lung DC, Yip CC, Cai JP, Chan JM, Chik TS, Lau DP, Choi CY, Chen LL, Chan WM, Chan KH, Ip JD, Ng AC, Poon RW, Luo CT, Cheng VC, Chan JF, Hung IF, Chen Z, Chen H, Yuen KY. Temporal profiles of viral load in posterior oropharyngeal saliva samples and serum antibody responses during infection by SARS-CoV-2: an observational cohort study. Lancet Infect Dis. 2020 May;20(5):565-574. doi: 10.1016/S1473-3099(20)30196-1. Epub 2020 Mar 23. PMID 32213337
- [Background] Luke TC, Casadevall A, Watowich SJ, Hoffman SL, Beigel JH, Burgess TH. Hark back: passive immunotherapy for influenza and other serious infections. Crit Care Med. 2010 Apr;38(4 Suppl):e66-73. doi: 10.1097/CCM.0b013e3181d44c1e. PMID 20154602
- [Background] Wong VW, Dai D, Wu AK, Sung JJ. Treatment of severe acute respiratory syndrome with convalescent plasma. Hong Kong Med J. 2003 Jun;9(3):199-201. PMID 12777656
- [Background] Kong LK, Zhou BP. Successful treatment of avian influenza with convalescent plasma. Hong Kong Med J. 2006 Dec;12(6):489. No abstract available. PMID 17148811
- [Background] Leider JP, Brunker PA, Ness PM. Convalescent transfusion for pandemic influenza: preparing blood banks for a new plasma product? Transfusion. 2010 Jun;50(6):1384-98. doi: 10.1111/j.1537-2995.2010.02590.x. Epub 2010 Feb 11. PMID 20158681
- [Background] Zhou B, Zhong N, Guan Y. Treatment with convalescent plasma for influenza A (H5N1) infection. N Engl J Med. 2007 Oct 4;357(14):1450-1. doi: 10.1056/NEJMc070359. No abstract available. PMID 17914053
- [Background] Wong HK, Lee CK, Hung IF, Leung JN, Hong J, Yuen KY, Lin CK. Practical limitations of convalescent plasma collection: a case scenario in pandemic preparation for influenza A (H1N1) infection. Transfusion. 2010 Sep;50(9):1967-71. doi: 10.1111/j.1537-2995.2010.02651.x. PMID 20412524
- [Background] Chen L, Xiong J, Bao L, Shi Y. Convalescent plasma as a potential therapy for COVID-19. Lancet Infect Dis. 2020 Apr;20(4):398-400. doi: 10.1016/S1473-3099(20)30141-9. Epub 2020 Feb 27. No abstract available. PMID 32113510
- [Background] Casadevall A, Pirofski LA. The convalescent sera option for containing COVID-19. J Clin Invest. 2020 Apr 1;130(4):1545-1548. doi: 10.1172/JCI138003. No abstract available. PMID 32167489
- [Background] Chang L, Yan Y, Wang L. Coronavirus Disease 2019: Coronaviruses and Blood Safety. Transfus Med Rev. 2020 Apr;34(2):75-80. doi: 10.1016/j.tmrv.2020.02.003. Epub 2020 Feb 21. PMID 32107119
- [Background] Hung IF, To KK, Lee CK, Lee KL, Chan K, Yan WW, Liu R, Watt CL, Chan WM, Lai KY, Koo CK, Buckley T, Chow FL, Wong KK, Chan HS, Ching CK, Tang BS, Lau CC, Li IW, Liu SH, Chan KH, Lin CK, Yuen KY. Convalescent plasma treatment reduced mortality in patients with severe pandemic influenza A (H1N1) 2009 virus infection. Clin Infect Dis. 2011 Feb 15;52(4):447-56. doi: 10.1093/cid/ciq106. Epub 2011 Jan 19. PMID 21248066
- [Background] Roback JD, Guarner J. Convalescent Plasma to Treat COVID-19: Possibilities and Challenges. JAMA. 2020 Apr 28;323(16):1561-1562. doi: 10.1001/jama.2020.4940. No abstract available. PMID 32219429
- [Background] Toy P. Update on transfusion-related acute lung injury. Clin Adv Hematol Oncol. 2019 Jul;17(7):378-381. No abstract available. PMID 31449502

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-06-25): https://cdn.clinicaltrials.gov/large-docs/09/NCT04468009/SAP_001.pdf
  • Informed Consent Form (2020-06-16): https://cdn.clinicaltrials.gov/large-docs/09/NCT04468009/ICF_000.pdf